CLINICAL TRIAL: NCT00973999
Title: A Randomised Placebo Controlled Trial to Explore the Effectiveness of Botulinum Toxin Injection at Reducing Oral Secretions and Frequency of Tracheal Suctioning in Tracheotomised Patients.
Brief Title: Botulinum Toxin and Saliva Management in Tracheotomised Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: HCA International Limited (Other)
Responsible Party: Mr. Chetan Vyas, HCA International Ltd.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CTO/09/032
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2009-09

CONDITIONS: Traumatic Brain Injury
Keywords: Botulinum Toxin; Saliva; Tracheostomy tube
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Botulinum Toxins; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Injection into salivary gland (Experimental)
  Interventions: Drug: Botulinum Toxin

INTERVENTIONS:
Drug: Botulinum Toxin — Each parotid salivary gland will be injected with 75MU of Botulinum Toxin type-A, 0.15mls in total, with 0.09mls into the mass of the gland and another 0.06mls into the adjacent part above the masseter muscle, using a 1ml syringe and a 30 gauge needle.
  Each submandibular salivary gland will be injected with 15MU of Botulinum Toxin A, administering 0.03mls, using a 1ml syringe and a 30 gauge needle.
  Other Names: Dysport, Ipsen Limited.

SUMMARY:
TITLE

A randomised placebo controlled trial to explore the effectiveness of Botulinum Toxin injection at reducing oral secretions and frequency of tracheal suctioning in tracheotomised patients.

DESIGN

Randomised controlled single blinded experimental design

AIMS

The purpose of this study is to determine if ultra-sounded guided injections of Botulinum Toxin into the salivary glands (Parotid and sub-mandibular glands) of patients with a tracheostomy tube in-situ assists in the reduction of oral secretions.

OUTCOME MEASURES

Amount of saliva production / frequency of tracheal suctioning / questionnaires.

POPULATION

In-patients at the Wellington Hospital based in London will be invited to participate within the study. Participants will be recruited from a range of wards which will include the Intensive Treatment Unit (ITU), acute medical wards and rehabilitation wards. All participants will have a tracheostomy tube in-situ and be breathing on room air, without the need for any mechanical ventilation. Participants will be receiving tracheal suctioning to assist in the clearance of saliva to maintain a clear airway.

A total of 40 participants will be recruited to the study across a two year period.

Each participant will have no prior history of the following:

* swallowing disorders
* stroke
* myocardial infarction
* head or neck surgery
* respiratory disease
* acute or progressive neurological disease
* structural abnormalities that could affect swallowing
* other medical conditions requiring medication that could affect swallowing.

ELIGIBILITY

Male and female adults over the age of 18 years

TREATMENT

Injection of Botulinum Toxin into both pairs of the parotid salivary glands and submandibular glands, using ultrasound guidance

DURATION

Data collection over a two year period / six weeks for each participant

DETAILED DESCRIPTION:
A randomised placebo controlled trial to explore the effectiveness of Botulinum Toxin injection at reducing oral secretions and frequency of tracheal suctioning in tracheotomised patients.

Protocol Number: Version 5, 20th July 2009

HCA reference: CTO/09/032

EudraCT reference: 2009-011204-27

This protocol describes the Botulinum toxin and Saliva management study and provides information about procedures for entering participants. Every care was taken in its drafting, but corrections or amendments may be necessary. These will be circulated to investigators in the study. Problems relating to this study should be referred, in the first instance, to the Chief Investigator. This study will adhere to the principles outlined in the NHS Research Governance Framework for Health and Social Care (2nd edition). It will be conducted in compliance with the protocol, the Data Protection Act and other regulatory requirements as appropriate

GLOSSARY OF ABBREVIATIONS

AE Adverse Event AR Adverse Reaction CTA Clinical Trials Authorisation CTO Clinical Trials Office CRF Case Report Form CRGO Clinical Research Governance Office MHRA Medicines and Healthcare Regulatory Agency REC Research Ethics Committee SAE Serious Adverse Event SUSAR Suspected Unexpected Serious Adverse Reaction

KEYWORDS Botulinum toxin, Saliva, Tracheostomy tube, Tracheal suctioning.

STUDY SUMMARY

TITLE A randomised placebo controlled trial to explore the effectiveness of Botulinum Toxin injection at reducing oral secretions and frequency of tracheal suctioning in tracheotomised patients.

DESIGN Randomised controlled single blinded experimental design AIMS The purpose of this study is to determine if ultra-sounded guided injections of Botulinum Toxin into the salivary glands (Parotid and sub-mandibular glands) of patients with a tracheostomy tube in-situ assists in the reduction of oral secretions.

OUTCOME MEASURES Amount of saliva production / frequency of tracheal suctioning / questionnaires.

POPULATION In-patients at the Wellington Hospital based in London will be invited to participate within the study. Participants will be recruited from a range of wards which will include the Intensive Treatment Unit (ITU), acute medical wards and rehabilitation wards. All participants will have a tracheostomy in-situ and be breathing on room air, without the need for any mechanical ventilation. Participants will be receiving tracheal suctioning to assist in the clearance of saliva to maintain a clear airway.

A total of 40 participants will be recruited to the study across a two year period.

Each participant will have no prior history of the following: (a) swallowing disorders; (b) stroke; (c) myocardial infarction; (d) head or neck surgery; (e) respiratory disease; (f) acute or progressive neurological disease; (g) structural abnormalities that could affect swallowing and (h) other medical conditions requiring medication that could affect swallowing.

ELIGIBILITY Adults over the age of 18 years

TREATMENT Injection of Botulinum toxin injections into both pairs of salivary glands (parotid and submandibular glands), using ultrasound guidance DURATION Data collection over a two year period / six weeks for each participant

1. INTRODUCTION

   1.1 BACKGROUND

   This Randomised Placebo Controlled trial will explore whether Botulinum Toxin injection into the salivary glands of tracheostomised patients is effective at reducing oral secretions and frequency of tracheal suctioning. The management of excess saliva ranges from conservative, such as postural changes and biofeedback to more aggressive such as medication, surgical and radiological intervention. Studies have shown that the use of medications, such as glycopyrrolate and scopolamine, are effective in reducing drooling, but have many adverse side effects, such as excessive dry mouth, constipation, urinary retention, decreased sweating and skin flushing 1-3. Recent research has shown that the long-term efficacy of intra-oral surgery for the management of sialorrhea to be minimally effective and that over two-thirds of patients had recurrence following surgery resulting in pharmacological or further surgical intervention 4. In contrast studies using radiation therapy in the management of sialorrhea, have shown initial satisfactory responses with up to 80% success rate, although there were some reported side effects, including oral candidiasis and mild skin reactions amongst participants 5

   Many studies have investigated the management of sialorrhea (drooling or excessive salivation) in both Parkinson's disease patients and in children with cerebral palsy, using Botulinum Toxin injected into the salivary glands 6-8. Several studies report on the use and efficacy of ultra-sound guided injection versus direct 'blind' injection into the salivary gland or glands 6 9-11, concluding that blind injections are as effective as ultra-sound guided injection, when solely injecting into the parotid gland. However, when injecting into both the parotid and submandibular glands use of guided injections as well as being a safe and effective technique in the treatment of sialorrhea 11 12. However to date there has been no application of Botulinum Toxin in patients who have a tracheostomy in-situ and who require regular tracheal suctioning due to excessive saliva and / or associated swallowing difficulties. This lack of knowledge may be of relevance given airway suctioning is associated with clinically significant complications, such as hypoxia microatelectasis (alveolar damage), laryngospasm and tracheal wall damage 13. Hooper suggested that the presence of a tracheostomy tube may cause irritation, resulting in an increased production of sputum 14.

   Patients have reported sensations of pain, pressure, crushing, choking and gagging, whereas in the hands of a skill practitioner, suctioning may not be more than a discomfort 15.

   Furthermore a study investigating knowledge and competence in performing tracheal suctioning in acute and within high dependency ward areas concluded that many staff members were unaware of recommended practice and a number demonstrated potentially unsafe practices 16.

   1.2 RATIONALE FOR CURRENT STUDY

   If ultra-sound guided Botulinum Toxin injection into the parotid and submandibular salivary glands is shown to be effective in reducing the amount of oral saliva and subsequently reducing for the need to perform tracheal suctioning, this can ultimately make tracheal suctioning unnecessary, reduce the time to extubation and normalise airflow through the larynx. This in turn may normalise swallowing physiology, with the ultimate outcome of removal of the tracheostomy tube.

   A reduction in salivary secretions may also significantly reduce the likelihood of aspiration pneumonia which may have a positive impact on length of stay as well as a reduction in healthcare costs.

   Given the wide-range of clinical competencies necessary for the safe and effective administration of tracheal suctioning, any pharmacologically induced benefit could attenuate the incidence of secondary complications as well as the likelihood of associated malpractice litigation.

   The current study will also aid in producing guidelines in the management of saliva in this patient population.
2. STUDY OBJECTIVES

   To determine whether Botulinum Toxin is effective at reducing oral secretions in tracheotomised patients.

   To determine whether Botulinum Toxin is effective at reducing the frequency of tracheal suctioning in tracheotomised patients.

   To investigate self-perceptions by patients in the management of oral / tracheal secretions

   To investigate nursing perceptions on amount oral secretions and frequency of tracheal suctioning
3. STUDY DESIGN

   The design will be a randomised, placebo-controlled single-blinded experimental study. Eligible patients will be randomly assigned to receive either active treatment or a placebo. Randomisation will be performed by matching consecutive eligible patients to a list of random numbers, generated via a computerised programme, allocating to either group.

   Each participant will be recruited for durations of six weeks in total. The treatment (injections of Botulinum toxin into the salivary glands) will be given one-week post after initial baseline measurements have been taken. Each participant will be followed-up at one week, two weeks and four weeks post injection. The patient will also continue to be reviewed throughout the study by the Speech and Language Therapist.

   3.1 STUDY OUTCOME MEASURES

   Primary Outcome measure

   To determine whether Botulinum Toxin is more effective than placebo at reducing oral secretions, as measured in milligrams at one week, two weeks and at four weeks follow up visits.

   Secondary Outcome measures

   To determine whether there is a difference in the frequency of tracheal suctioning performed, across a 12-hour period, between the treatment and placebo controlled group, as measured by the volume of secretions suctioned at one week, two weeks and four weeks follow up visits.

   To investigate the self-perceived patient outcomes of amount of oral secretions and frequency of tracheal suctioning required, using a self-perception questionnaire, to be completed at one week, two weeks and at four weeks follow up visits.

   To investigate nursing perceptions on the amount of oral secretions and frequency tracheal suctioning required by individual patients, using a questionnaire, to be completed at one week, two weeks and at four weeks follow up visits.
4. PARTICIPANT ENTRY

   4.1 PRE-RANDOMISATION EVALUATIONS

   All participants will be referred to the speech and language therapy department by their primary Consultant, for assessment of their tracheostomy, communication and / or swallowing.

   The patient will be assessed by the Speech and Language Therapist, using a Clinical Bedside Evaluation (CBE), as to whether they are able to safely swallow their own saliva or require tracheal suctioning to assist in clearing secretions that are falling into their airway.

   4.2 INCLUSION CRITERIA

   Patients must meet all of the following inclusion criteria to be eligible for enrolment into the study;

   Male or female participants over the age of 18 years

   Participants who have a tracheostomy tube in-situ

   Participants who are breathing on room air, without the need for any mechanical ventilation

   Participants who require tracheal suctioning in order to maintain a clear airway

   4.3 EXCLUSION CRITERIA

   Patients presenting with any of the following exclusion criteria will not be included in the study;

   Contra-indications to the use of Botulinum Toxin

   Receiving medications that may react with Botulinum Toxin, such as aminoglycosides (e.g., gentamicin), anticholinesterase medicines (e.g., neostigmine), lincosamides (e.g., clindamycin), magnesium, neuromuscular blockers (e.g., atracurium), polymyxin, or quinidine because the risk of toxic effects may be increased

   Receiving anticoagulants medication (e.g., warfarin)

   Expectant mothers

   Previous history of;

   Swallowing disorders Stroke Myocardial Infarction Heart Disease Head or neck surgery Acute or progressive neurological disease Structural abnormalities that may affect swallowing

   4.4 WITHDRAWAL CRITERIA

   Patients will be able to withdraw from the study at any time and will continue to receive therapy intervention / treatment as is required. Subjects may be withdrawn from the study for any of the following reasons;

   Personal reasons: as stated in the informed consent form, subjects may withdraw from the study at any time

   Subject withdraws consent

   Clinical judgement of the Investigator: a subject may be withdrawn from the study, if the opinion of the Investigator, it is not in the subject's best interest to continue

   Loss to follow-up

   If the patient withdraws from the study and also withdraws consent for disclosure of future information, no further evaluations will be performed and no additional data collected. The investigator will retain and continue to use any data collected before such withdrawal of consent.

   Withdrawal due to an adverse event should be distinguished from that due to patient perceived lack of treatment response or any other reason for withdrawal and recorded on the appropriate adverse event Case Report Form.

   If a patient withdraws due to a serious adverse event, the serious adverse event will be reported in accordance with the reporting requirements defined in Section 7, Pharmacovigilence.
5. RANDOMISATION AND ENROLMENT PROCEDURE

   5.1 RANDOMISATION OR REGISTRATION PRACTICALITIES

   From the 40 participants who will be enrolled within the study, 20 will be randomly assigned to the treatment group and the other 20 will be randomly allocated to the placebo-control group.

   All participants will be randomised to either the treatment or placebo-controlled group using a computerised randomisation generator (www.Randomization.com). This process will be co-ordinated by the CTO administrator who will advise the Chief Investigator to which group consecutive participants are allocated.

   5.2 UNBLINDING

   All participants and Nursing staff will be blinded to which group each participant has been allocated to. In the event where patients become unwell during the study or where there is a SAE, where the treatment would affect future management, unblinding will occur and all parties involved in the participants care will be informed as to which group the participant was allocated, as well as informing the patient and their carers.
6. TREATMENTS

   Dr. V P Misra, Consultant Neurophysiologist, will be responsible for prescribing the study medication, for patients receiving the Botulinum Toxin within the treatment arm of the study.

   6.1 TREATMENT ARMS

   The dosage given is as follows:

   Botulinum Toxin type-A (Dysport, Ipsen Ltd, Slough, Berkshire) will be reconstituted with 1.0ml of sodium chloride injection B.P. (0.9%) to yield a solution containing 500 units per ml of Dysport.

   Each parotid salivary gland will be injected with 75MU of Botulinum Toxin type-A (Dysport, Ipsen Ltd, Slough, Berkshire), 0.15mls in total, with 0.09mls into the mass of the gland and another 0.06mls into the adjacent part above the masseter muscle, as described by Pal 17, using a 1ml syringe and a 30 gauge needle.

   Each submandibular salivary gland will be injected with 15MU of Botulinum Toxin A (Dysport, Ipsen Ltd, Slough, Berkshire), administering 0.03mls, using a 1ml syringe and a 30 gauge needle.

   Each injection will be performed using ultrasound guidance using the Philips iU22 ultrasound system to landmark the site of each of the glands. The drug will be obtained from Ipsen Ltd and funding application for the drug will be made to Ipsen Ltd, as well as via The Wellington Hospital.

   Placebo Participants will receive a pin-pick using a 1ml syringe and a 30 gauge needle, filled with sodium chloride (0.9%) at the sites of the parotid and submandibular salivary glands, using ultrasound guidance to landmark the sites.

   6.2 INTERACTION WITH OTHER DRUGS

   According to the summary of product characteristics produced by Ipsen limited, drugs which affect neuromuscular transmission, such as aminoglycoside antibiotics, should be used with caution. Other medications that may interact with Botulinum Toxin are anticholinesterase medicines (e.g., neostigmine), lincosamides (e.g., clindamycin), magnesium, neuromuscular blockers (e.g., atracurium), polymyxin, or quinidine because the risk of toxic effects may be increased.

   6.3 DISPENSING AND ACCOUNTABILITY

   The shelf-life of Botulinum toxin- type A is 15 months, when stored at a temperature of 2-8oC. The product can be stored for up to 8 hours, following reconstitution at a temperature of 2-8oC. The drug will be stored with the Wellington Hospitals Pharmacy department and be prepared by the Consultant Neurophysiologist prior to administration. Once used, any remaining Botulinum Toxin will be inactivated with dilute hypochlorite solution and thereafter be disposed of using the hospitals' policy on disposal of unused drugs; any out-of-date vials of the drug will also be inactivated with dilute hypochlorite and disposed using the hospitals practice policy on disposal of medication / drugs.
7. PHARMACOVIGILANCE

   7.1 DEFINITIONS

   Adverse Event (AE):

   Any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational medicinal product (IMP), whether or not considered related to the IMP.

   Adverse Reaction (AR):

   All untoward and unintended responses to an IMP related to any dose administered. All AEs judged by either the reporting investigator or the sponsor as having reasonable causal relationship to a medicinal product qualify as adverse reactions. The expression reasonable causal relationship means to convey in general that there is evidence or argument to suggest a causal relationship.

   Unexpected Adverse Reaction: an AR, the nature or severity of which is not consistent with the applicable product information (e.g. investigator's brochure for an unapproved investigational product or summary of product characteristics (SmPC) for an authorised product). When the outcome of the adverse reaction is not consistent with the applicable product information this adverse reaction should be considered as unexpected. Side effects documented in the SmPC which occur in a more severe form than anticipated are also considered to be unexpected.

   Serious Adverse Event (SAE) or Serious Adverse Reaction:

   Any untoward medical occurrence or effect that at any dose Results in death

   Is life-threatening - refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe

   Requires hospitalisation, or prolongation of existing inpatients' hospitalisation

   Results in persistent or significant disability or incapacity

   Is a congenital anomaly or birth defect

   Medical judgement should be exercised in deciding whether an AE/AR is serious in other situations. Important AE/ARs that are not immediately life-threatening or do not result in death or hospitalisation but may jeopardise the subject or may require intervention to prevent one of the other outcomes listed in the definition above, should also be considered serious.

   Suspected Unexpected Serious Adverse Reaction (SUSAR):

   Any suspected adverse reaction related to an IMP that is both unexpected and serious.

   7.2 CAUSALITY

   Most adverse events and adverse drug reactions that occur in this study, whether they are serious or not, will be expected treatment-related toxicities due to the drugs used in this study. The assignment of the causality should be made by the investigator responsible for the care of the participant using the definitions in the table below.

   If any doubt about the causality exists the local investigator should inform the study coordination centre who will notify the Chief Investigators. The pharmaceutical companies and/or other clinicians may be asked to advise in some cases.

   In the case of discrepant views on causality between the investigator and others, all parties will discuss the case. In the event that no agreement is made, the MHRA will be informed of both points of view.

   Relationship Description Unrelated There is no evidence of any causal relationship Unlikely There is little evidence to suggest there is a causal relationship (e.g. the event did not occur within a reasonable time after administration of the trial medication). There is another reasonable explanation for the event (e.g. the participant's clinical condition, other concomitant treatment).

   Possible There is some evidence to suggest a causal relationship (e.g. because the event occurs within a reasonable time after administration of the trial medication). However, the influence of other factors may have contributed to the event (e.g. the participant's clinical condition, other concomitant treatments).

   Probable There is evidence to suggest a causal relationship and the influence of other factors is unlikely.

   Definitely There is clear evidence to suggest a causal relationship and other possible contributing factors can be ruled out.

   Not assessable There is insufficient or incomplete evidence to make a clinical judgement of the causal relationship.

   7.3 REPORTING PROCEDURES

   All adverse events will be reported. Depending on the nature of the event the reporting procedures below should be followed. Any questions concerning adverse event reporting should be directed to the study coordination centre in the first instance. A flowchart is given below to aid in the reporting procedures.

   7.3.1 Non serious AR / AEs

   All such toxicities, whether expected or not, will be recorded in the toxicity section of the relevant case report form and sent to the study coordination centre within one month of the form being due.

   7.3.2 Serious AR / AEs

   Fatal or life threatening SAEs and SUSARs will be reported on the day that the local site is aware of the event. The SAE form asks for nature of event, date of onset, severity, corrective therapies given, outcome and causality (i.e. unrelated, unlikely, possible, probably, definitely). The responsible investigator should sign the causality of the event. Additional information should be sent within 5 days if the reaction has not resolved at the time of reporting.

   SAEs

   An SAE form should be completed and faxed to the study coordination centre for all SAEs within 24 hours. Please refer to the product SMPC for details of adverse events, if not included within these guidelines then any adverse effects will be reported to the Clinical Trials Office

   SUSARs

   In the case of serious, unexpected and related adverse events, the staff at the site should:

   Complete the SAE case report form & send it immediately (within 24 hours, preferably by fax), signed and dated to the study coordination centre together with relevant treatment forms and anonymised copies of all relevant investigations.

   Or

   Contact the study coordination centre by phone and then send the completed SAE form to the study coordination centre within the following 24 hours as above.

   The study coordination centre will notify the MHRA and REC of all SUSARs occurring during the study according to the following timelines; fatal and life-threatening within 7 days of notification and non-life threatening within 15 days. All investigators will be informed of all SUSARs occurring throughout the study.

   Local investigators should report any SUSARs and /or SAEs as required by their Local Research Ethics Committee and/or Research & Development Office.

   Contact details for reporting SAEs and SUSARs

   Fax: 020 7034 8402, for the immediate attention Rasmi Pillai

   Please send SAE forms to:

   Rasmi Pillai 79 Harley Street London W1G 8PZ

   Tel: 0207 034 8403 (Mon to Fri 09:00 - 17:00 hours)
8. ASSESSMENT AND FOLLOW-UP

   Participants will continue to be followed-up at one week, two week and at four week intervals post intervention and thereafter as long as they have their tracheostomy tube in-place and continue to benefit from ongoing intervention from Speech and Language Therapy for swallowing and / or communication difficulties. Assessment will focus on weaning from the tracheostomy tube, ability to safely swallow and recordings of tracheal suctioning and amount of oral saliva. Assessments will also be made of the patients / carers perceptions of saliva management.

   8.1 LOSS TO FOLLOW-UP

   Patients who may be lost to follow-up will not have their data included and will be followed-up locally by their local services.

   8.2 TRIAL CLOSURE

   Participants will continue to receive Speech and Language Therapy intervention and ongoing assessment, whilst they remain an inpatient at the hospital. They will be removed from the trial if and when they are swallowing and managing their own saliva, without any need for any tracheal suctioning and if the tracheostomy tube is removed. The end of trial date will be six weeks from inclusion date.
9. STATISTICS AND DATA ANALYSIS

   A power calculation has been performed to determine the sample size, which has been based on previous studies using Botulinum Toxin type A and treatment of drooling / excessive saliva management.

   Once entered into Statistical Package for the Social Sciences (SPSS) the data will be examined for extreme values and transcription errors. Data analysis will commence following data base lock, which will occur four to six weeks following the last patient data collection and resolution of all outstanding data queries. Data will be analysed using Multiple Regression.

   Data and all appropriate documentation will be stored for a minimum of 5 years after the completion of the study, including the follow-up period.
10. MONITORING

    10.1 RISK ASSESSMENT

    This study is considered low risk as this drug dosage has been shown to be a safe and effective treatment for Parkinson's disease patients with excess saliva (sialorrhea).

    10.2 MONITORING AT STUDY COORDINATION CENTRE

    During study conduct, HCA's CTO will conduct periodic monitoring visits to the investigator site to ensure that the protocol and GCP are being followed. The monitors may review source documents to confirm that the data recorded on the CRF is accurate. The investigator and institution will allow HCA' CTO and appropriate regulatory authorities direct access to source documents to perform this verification.

    The study site may be subject to quality assurance audits performed by HCA's CTO.

    It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and audits or inspections and that sufficient time is devoted to the process.
11. REGULATORY ISSUES

    11.1 CTA

    This study is being conducted under a Clinical Trial Authorisation issued by the UK Competent Authority; the Medicines and Healthcare products Regulatory Agency (MHRA); EudraCT No. 2009-011204-2742

    11.2 ETHICS APPROVAL

    This protocol will be submitted to the Ethics Committee (EC), whose approval will be obtained before the start of the study. The investigators will inform the EC of subsequent protocol amendments and any serious adverse events which occur during the study.

    11.3 CONSENT

    THE INVESTIGATOR OR DELEGATED PHYSICIAN MUST INFORM PATIENTS ABOUT THE BACKGROUND TO, AND PRESENT KNOWLEDGE OF THE IMP WITH SPECIAL REFERENCE TO KNOWN ACTIVITY AND ADVERSE DRUG REACTION. THE INVESTIGATORS MUST ALSO ENSURE THE FOLLOWING POINTS ARE MADE:

    The patient must be provided with the Patient Information Sheet and Informed Consent form consistent with the protocol version used and approved by EC.

    Before the patient is entered into the study, the patient's written consent must be obtained using the Informed Consent form described above (according to HCA SOP RD.CTS.UK.001). The patient will retain a copy of the signed informed consent form and the original will be filed in the Trial Master file.

    The patient may refuse treatment either before or at any time during the study. Refusal to participate will involve no penalty or loss of benefits to which the patient is otherwise entitled.

    An explanation on whom to contact for answers to pertinent questions about the research and research subject's rights, and who to contact in the event of a research-related injury to the subject must be given.

    All participants are free to withdraw at any time from the protocol treatment without giving reasons and without prejudicing further treatment.

    11.4 CONFIDENTIALITY

    Participants' identification data will be required for the registration process. The Study Coordination Centre will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act.

    11.5 INDEMNITY

    HCA International Ltd. holds negligent harm insurance policies which apply to this study.

    11.6 SPONSOR

    HCA International Ltd, The Clinical Trials Office will act as the main sponsor for this study.

    11.7 FUNDING

    HCA International Ltd

    11.8 AUDITS AND INSPECTIONS

    The study may be subject to inspection and audit by HCA international. Under their remit as a Department of Health recognised Sponsor HCA will ensure adherence to GCP and the Research Governance Framework for Health and Social Care (2nd edition). The study will be monitored for Research Governance compliance in accordance with HCA SOP No RD.RG.UK.001.
12. STUDY MANAGEMENT

The day-to-day management of the study will be co-ordinated through the Clinical Trials Office.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study
* Male or female participants over the age of 18 years
* Participants who have a tracheostomy tube in-situ
* Participants who are breathing on room air, without the need for any mechanical ventilation
* Participants who require tracheal suctioning in order to maintain a clear airway

Exclusion Criteria:

* Patients presenting with any of the following exclusion criteria will not be included in the study
* Contra-indications to the use of Botulinum Toxin
* Receiving medications that may react with Botulinum Toxin, such as aminoglycosides (e.g., gentamicin), anticholinesterase medicines (e.g., neostigmine), lincosamides (e.g., clindamycin), magnesium, neuromuscular blockers (e.g., atracurium), polymyxin, or quinidine because the risk of toxic effects may be increased
* Receiving anticoagulants medication (e.g., warfarin)
* Expectant mothers
* Previous history of:

  * Swallowing disorders
  * Stroke
  * Myocardial Infarction
  * Heart Disease
  * Head or neck surgery
  * Acute or progressive neurological disease
  * Structural abnormalities that may affect swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
The weight of intra-orally placed dental rolls | participants will be followed for the duration of hospital stay, an expected average of 12 weeks

SECONDARY OUTCOMES:
Observational tally of number of tracheal suctions performed over a 12-hour period. | participants will be followed for the duration of hospital stay, an expected average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chetan Vyas, BSc, MSc, Principal Investigator — HCA International Limited
Locations (1):
- The Wellington Hospital, London, United Kingdom